CLINICAL TRIAL: NCT05211557
Title: A Single-Arm, Open-Label Study to Evaluate Safety and Efficacy of Fully Human B7H3 CAR-T in Treating Patients With Recurrent Malignant Ovarian Cancer
Brief Title: Study of Fully Human B7H3 CAR-T in Treating Recurrent Malignant Ovarian Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Collaborators: Xuzhou Medical University (Other); IIT MediTech (Jiangsu) Co. Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2021-KL184-01
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Ovarian Cancer
Keywords: Fully Human B7H3 CAR-T; Recurrent Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fhB7H3.CAR-T cells (Experimental): In phase I study, 9 enrolled patients diagnosed with advanced ovarian cancer will receive one-time infusion of fhB7H3.CAR-Ts at the doses of 1×10^6/kg, 3×10^6/kg and 5×10^6/kg, 3 patients for each dose. To further confirm the therapeutic efficacy, in phase II study, 6 enrolled patients will receive an optimal dose (balancing effectiveness and toxicity) of fhB7H3.CAR-Ts. Prior to receiving the infusions, patients will undergo lymphodepletion with fludarabine and cyclophosphamide.
  Interventions: Biological: fhB7H3.CAR-Ts

INTERVENTIONS:
Biological: fhB7H3.CAR-Ts — Three dose levels will be evaluated: Dose Level 1 (1×10^6/kg), dose Level 2 (3×10^6/kg) and dose Level 3 (5×10^6/kg). If dose limiting toxicities (DLTs) are observed in each doses, Dose Level -1 (0.5×10^6/kg /infusion) will be evaluated.
  Other Name: B7H3 targeting chimeric antigen receptor T cells Drug: Fludarabine 30 mg/m2 i.v. for 3 consecutive days (Day -5~Day -3) Other Name: FLUDARA Drug: Cyclophosphamide 750 mg/m2 i.v. for once (Day -5) Other Name: Cytoxan

SUMMARY:
This is single center, open-label phase I, non-randomized study which will enroll patients with recurrent advanced ovarian cancer to evaluate the safety, feasibility, and efficacy of fully human B7H3 CAR-T cells (fhB7H3.CAR-Ts) via using a '3+3+3' dose escalation design. In the dose expansion cohort, six patients will be enrolled to further assess their efficacy with the optimal dosage.

DETAILED DESCRIPTION:
The purpose of this study is to test the safety and efficacy of a newly developed fully human scFv-armed B7H3 targeting chimeric antigen receptor T cells (fhB7H3.CAR-Ts), which are supposed to attack and eliminate B7H3-positive cancer cells. The patients who have been diagnosed as recurrent or relapsed malignant ovarian cancer, especially ovarian cancer patients with refractory ascites, will be potentially enrolled after assessing the expression of B7H3 antigen in tumor tissue by immunohistochemistry staining or ascitic tumor cells by flow cytometry.

After enrollment, participants' peripheral blood mononuclear cells will be collected and used to manufacture fhB7H3.CAR-Ts. Before infusion, the patients will receive lymphodepletion chemotherapy with cyclophosphamide and fludarabine for three consecutive days. Two days later after lymphodepletion, the fhB7H3.CAR-Ts would be given through an abdominal catheter for intraperitoneal infusion. From the day of infusion, participants' peripheral blood and ascites will be collected twice a week in the first month for monitoring the survival of fhB7H3.CAR-Ts and evaluating the therapeutic efficacy. Additional follow-up and examination will be performed monthly for the first three month and then trimonthly until one year. Thereafter, annual follow-up will be completed for 5 years.

In addition, since the fhB7H3.CAR-Ts containing a RQR8 safety-switch which could be targeted and removed by Rituximab. Participants who experience life-threatening toxicities caused by uncontrollable proliferation of fhB7H3.CAR-Ts will receive infusion of Rituximab (Rituxan or Ruxience or Halpryza) to assess the ability of RQR8 safety-switch to eliminate infused fhB7H3.CAR-Ts.

This is an investigator-initiated clinical study to assess first-line clinical performance of novel fhB7H3.CAR-Ts which may help other advanced and recurrent ovarian cancer patients in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Procurement and T-cell production eligibility: a previously evaluation confirmed autologous peripheral blood mononuclear cells can be used for T-cell production
2. Written informed consent and authorization for release of personal health information
3. Subject has adequate performance status as defined by ECOG score of ≤ 2.
4. Expected life expectancy is no less than 12 weeks.
5. Subjects must have histologically or cytologically confirmed ovarian cancer. And cancer tissue or ascitic cancer cells are measured positive for B7H3 expression.
6. Subjects must have recurrent or refractory disease after or during first-line treatment.

   Defined as:

   Radiographic progression or Continuous Elevation of CA125.
7. Subjects must have evaluable disease - defined as:

   Measurable disease with tumor length ≥ 10mm or enlarged lymph nodes ≥ 15mm according to RECIST v1.1 criteria.
8. Adequate organ function - defined as:

   1. Blood routine:

      white blood cell count ≥ 3 × 10^9 / L; neutrophil count ≥ 1.5 × 10^9 / L; hemoglobin ≥ 9g/dL; platelet count ≥ 80 × 10^9 / L; INR< 1.5 × ULN; PT, APTT< 1.5 × ULN
   2. The liver, kidney, lung and cardiopulmonary function:

   Urea and serum creatinine ≤ 1.5 × ULN; Left ventricular ejection fraction ≥ 40%; Baseline oxygen saturation ≥ 95%; Total bilirubin ≤ 1.5 × ULN; ALT and AST ≤ 3 × ULN.
9. Not pregnant with negative serum pregnancy test within 3 days prior to enrollment.
10. Female subjects of childbearing potential must be willing to abstain from heterosexual activity or to use 2 forms of highly effective methods of contraception from the time of informed consent until 8 weeks after study treatment discontinuation.

    -

Exclusion Criteria:

1. Subject has primary immunodeficiency syndrome or history of severe allergic reaction.
2. Subject has active infection with HIV, HTLV, HBV, HCV.
3. Subject has severe, uncontrolled intercurrent bacterial, viral or fungal infection.
4. Subject has a history of gastrointestinal perforation, clinical and/or radiographic evidence of bowel obstruction, or intra-abdominal abscess within 3 months prior to starting treatment.
5. Subject has active malignancy under treatment other than ovarian cancer.
6. Subject has Grade ≥ 3 cardiac dysfunction or symptomatic arrhythmia requiring intervention.
7. Subject is current using of systemic corticosteroids at doses ≥10 mg prednisone daily or its equivalent.
8. Subject has not recovered from toxicity of previous anti-tumor treatment (CTCAE 5.0).
9. Subject is pregnant or breastfeeding.
10. Unwilling or unable to provide consent/assent for participation in the study. -

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity of fully human B7H3 CAR-T cells | 1 month
  Dose limiting toxicity (DLT), including the type, frequency, severity and duration of adverse events, such as cytokine release syndrome (CRS), on-target off-tumor, immune effector cell-associated neurotoxicity syndrome, will be monitored and assessed.
Objective response of fully human B7H3 CAR-T cells | 1 month
  Objective response rate (ORR) including complete response (CR), partial response (PR), and/or stable disease, will be determined by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
  Complete Response (CR): disappearance of all target lesions. Partial Response (PR): >=30% decrease in the sum of the longest diameter of target lesions. Stable Disease (SD): no response or less response than Partial or Progressive.
  Progressive Disease (PD): 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.

SECONDARY OUTCOMES:
In vivo persistence of fully human B7H3 CAR-T cells | 1 month
  Presence and number of CAR T cells in the peripheral blood and ascites will be assessed.

OTHER OUTCOMES:
Progress free survival (PFS) | up to 5 years
  PFS will be assessed from the time of lymphodepletion prior to infusion of fhB7H3.CAR-Ts to
Overall survival (OS) | up to 5 years
  OS will be assessed from the date of lymphodepletion prior to infusion of fhB7H3.CAR-Ts to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Junnian Zheng, M.D., Ph.D., Study Director — The Affiliated Hospital of Xuzhou Medical University, Xuzhou Medical University; Longzhen Zhang, M.D., Ph.D., Principal Investigator — The Affiliated Hospital of Xuzhou Medical University; Gang Wang, Ph.D., Principal Investigator — Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No